CLINICAL TRIAL: NCT02365142
Title: Phase I/II. Treatment of Osteoarthritis by Intra-articular Injection of Bone Marrow Mesenchymal Stem Cells With Platelet Rich Plasma(PRGF)
Brief Title: Treatment of Osteoarthritis by Intra-articular Injection of Bone Marrow Mesenchymal Stem Cells With Platelet Rich Plasma
Acronym: CMM-PRGF/ART
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CMM-PRGF/ART; 2011-006036-23 (EudraCT Number)
Record Dates: First submitted 2014-07-18; First posted 2015-02-18 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Mesenchimal stem cell; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet Rich Plasma (PRGF) (Active Comparator): Platelet Rich plasma (PRGF) 3 intraarticular onjections sepataded by 7 days.
  Interventions: Biological: Platelet Rich plasma (PRGF)
- BMMSC with Platelet Rich Plasma (PRGF) (Active Comparator): Single intraarticular injection of 100 million Bone marrow mesenchimal stem cells and three intraarticular injections of plateler Rich Plasma (PRGF) separatede by 7 days.
  Interventions: Biological: 100 million Bone marrow mesenchimal stem cells; Biological: Platelet Rich plasma (PRGF)

INTERVENTIONS:
Biological: 100 million Bone marrow mesenchimal stem cells — 100 million Bone marrow mesenchimal stem cells with PRGF
  Arms: BMMSC with Platelet Rich Plasma (PRGF)
Biological: Platelet Rich plasma (PRGF) — 3 injections of PRGF

SUMMARY:
Purpose: To determine the safety, feasibility and effectiveness (clinical and radiological) of intra-articular administration of autologous mesenchymal stem cells (MSCs) with platelet richa plasma (PRGF) in patients with knee osteoarthritis.

Patients and methods

Clinical trial phase I- II, randomized , multicenter , with two treatment arms and 19 patients for each group. The investigators compare the intraarticular injection of against the administration of two different doses of mesenchymal stem cells with hialuronic acid according to the following scheme:

1. Group A: 3 intra-articular injections of platelet rich plasma (PRGF®) separated by 7 days.
2. Group B: 3 intra-articular injections of platelet richa plasma (PRGF®) separated by 7 days and one with Mesenchimal stems cells. Intra-articular injection of 100 million autologous mesenchymal progenitor stem cells cultured ex - vivo (cell suspension sterile small volume (5-10 ml ) in a vehicle suitable for intraarticular injection ) followed by an intraarticular injection of platelet richa plasma (PRGF®). The treatment is completed with 2 more injection of platelet richa plasma (PRGF®) separeted by one week.

In addition the investigators assess the response to intra-articular infusion of CMM analyzing the following parameters:

* Clinical assessment of pain and function (Baseline, 1, 3, 6 and 12 months since treatment): VAS , WOMAC , KOOS , EuroQol, SF-16, Lequesne , WOMAC , KOOS.
* Radiographic (baseline and 12 months from treatment): Femorotibial space.
* Radiographic using MRI (baseline and 12 months from treatment): by assessing the number location of the lesions , cartilage thickness , signal intensity , subchondral bone alteration , volume and WORMS and dGEMRIC protocols.

DETAILED DESCRIPTION:
Purpose: To determine the safety, feasibility and effectiveness (clinical and radiological) of intra-articular administration of autologous mesenchymal stem cells (MSCs) with platelet richa plasma (PRGF®) in patients with knee osteoarthritis.

Patients and methods

Clinical trial phase I- II, randomized , multicenter , with two treatment arms and 19 patients for each group. The investigators compare the intraarticular injection of against the administration of two different doses of mesenchymal stem cells with hialuronic acid according to the following scheme:

1. Group A: 3 intra-articular injections of platelet richa plasma (PRGF®) separated by 7 days.
2. Group B: 3 intra-articular injections of platelet richa plasma (PRGF®) separated by 7 days and one with Mesenchimal stem cell. Intra-articular injection of 100 million autologous mesenchymal progenitor stem cells cultured ex - vivo (cell suspension sterile small volume (5-10 ml ) in a vehicle suitable for intraarticular injection ) followed by an intraarticular injection of platelet richa plasma (PRGF®). The treatment is completed with 2 more injection of platelet richa plasma (PRGF®) separeted by one week.

The autologous mesenchymal stem cells are obtained from the iliac crest under local anesthesia and sedation. They are cultured ex vivo The primary endpoint is safety and feasibility. The investigators registered the occurrence of complications and / or adverse effects during the study.

In addition the investigators assess the response to intra-articular infusion of CMM analyzing the following parameters:

* Clinical assessment of pain and function (Baseline, 1, 3, 6 and 12 months since treatment): VAS , WOMAC , KOOS , EuroQol, SF-16, Lequesne , WOMAC , KOOS.
* Radiographic (baseline, 6 and 12 months since treatment): Femorotibial space.
* Radiographic using MRI (baseline, 6 and 12 months since treatment): by assessing the number location of the lesions , cartilage thickness , signal intensity , subchondral bone alteration , volume and WORMS and dGEMRIC protocols.

All patients met the following inclusion and exclusion criteria:

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 40 and 80 year old
* Bad results with previous hyaluronic acid injection
* Diagnosis of knee OA according to the criteria of osteoarthritis of the ACR (American College of Rheumatology)
* Joint pain equal or greater than 2.5 points on the visual analogue scale (VAS)
* Radiological Classification: Kellgren-Lawrence scale greater or equal to 2
* Body mass index between 20 and 35 kg/m2
* Ability to follow during the study period

Exclusion Criteria:

* Bilateral Osteoarthritis of the Knee requiring treatment in both knees
* Previous diagnosis of polyarticular disease
* Severe mechanical deformation
* Arthroscopy during the previous 6 months
* Intraarticular infiltration of hyaluronic acid in the last 6 months
* Systemic autoimmune rheumatic disease
* Poorly controlled diabetes mellitus
* Blood dyscrasias
* Immunosuppressive or anticoagulant treatments
* Treatment with corticosteroids in the 3 months prior to inclusion in the study
* NSAID therapy within 15 days prior to inclusion in the study
* Patients with a history of allergy to penicillin or streptomycin

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Baseline Visual analogue scale (VAS) Baseline Visual analogue scale (VAS) | Day 1
  Baseline Visual analogue scale (VAS) prior to the initial dose on day 1
Baseline value of knee injury and osteoarthritis outcome score (Koos). | Day 1
  Prior to the intervention on day 1 value of knee injury and osteoarthritis outcome score (Koos).
Baseline Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC). | Day 1
  Universities Osteoarthritis Index score (WOMAC).
Baseline SF-36 value | Day 1
  Baseline SF-36 value
Baseline euroquol 5D value | Day 1
  Pretreatment euroquol 5D value
Baseline Lequesne index | Day 1
  Prior to the intervention on day 1 Lequesne index
Baseline femorotibial distance | Day 1
  Prior to the intervention femoritibial distance on rosenberg x-ray view
Number of Participants with Serious and Non-Serious Adverse Events Number of Participants with Serious and Non-Serious Adverse Events Number of Participants with Serious and Non-Serious Adverse Events | Follow up (up to 12 months)
  Participants with Serious and Non-Serious Adverse Events Number of Participants with Serious and Non-Serious Adverse Events During the follow up
Visual analogue scale (VAS) at 1 month | 1 month
  Visual analogue scale (VAS) at on month
Visual analogue scale (VAS) at 3 months | 3 months
  Visual analogue scale (VAS) at 3 months
Visual analogue scale (VAS) at 6 months | 6 months
  Visual analogue scale (VAS) at 6 months
Visual analogue scale (VAS) at 12 months | 12 months
  Visual analogue scale (VAS) at 12 months
Value of knee injury and osteoarthritis outcome score (Koos) at 1 month | 1 month
  Value of knee injury and osteoarthritis outcome score (Koos) at 1 month
Value of knee injury and osteoarthritis outcome score (Koos) at 3 month | 3 Months
  Value of knee injury and osteoarthritis outcome score (Koos) at 3 month
Value of knee injury and osteoarthritis outcome score (Koos) at 6 month | 6 months
  Value of knee injury and osteoarthritis outcome score (Koos) at 6 month
Value of knee injury and osteoarthritis outcome score (Koos) at 12 months | 12 months
  Value of knee injury and osteoarthritis outcome score (Koos) at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: José Lamo-Espinosa, MD, Principal Investigator — Clinica Universidad de Navarra; Felipe Prosper, MD, PhD, Study Director — Clínica Universidad de Navarra; Juan Blanco, MD; PhD, Principal Investigator — Complejo Universitario de Salamanca
Locations (2):
- Spain (2):
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Departamento Cirugía Ortopédica y Traumatología. Clinica Universidad de Navarra, Pamplona, Navarre

REFERENCES:
- [Derived] Lamo-Espinosa JM, Blanco JF, Sanchez M, Moreno V, Granero-Molto F, Sanchez-Guijo F, Crespo-Cullel I, Mora G, San Vicente DD, Pompei-Fernandez O, Aquerreta JD, Nunez-Cordoba JM, Vitoria Sola M, Valenti-Azcarate A, Andreu EJ, Del Consuelo Del Canizo M, Valenti-Nin JR, Prosper F. Phase II multicenter randomized controlled clinical trial on the efficacy of intra-articular injection of autologous bone marrow mesenchymal stem cells with platelet rich plasma for the treatment of knee osteoarthritis. J Transl Med. 2020 Sep 18;18(1):356. doi: 10.1186/s12967-020-02530-6. PMID 32948200
- See also: University clinic of navarre trial information — http://www.cun.es/actualidad/noticias/celulas-madre-osea-artrosis-rodilla